CLINICAL TRIAL: NCT01603069
Title: A Phase IIa, 12 Week, Multicentre, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Assess the Safety and Tolerability of Oral AZD3241 in Patients With Parkinson's Disease
Brief Title: A Study to Assess Safety and Tolerability of Oral AZD3241 in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0490C00005; EudraCT number: 2012-001313-16
Record Dates: First submitted 2012-05-14; First posted 2012-05-22 (Estimated); Last update posted 2013-07-19 (Estimated); Status verified 2013-07

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Safety; Tolerability
MeSH Terms: conditions — Parkinson Disease | interventions — AZD3241; BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- AZD3241, 300 mg (Active Comparator): AZD3241 300 mg BID
  Interventions: Drug: AZD3241 300 mg BID
- AZD3241, 600 mg (Active Comparator): AZD3241 600 mg BID
  Interventions: Drug: AZD3241 600 mg BID
- Placebo (Placebo Comparator): Placebo to AZD3241
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3241 300 mg BID — The following dose escalation schedule will be used for 300 mg BID: 100 mg BID from Day 1 through Day 7. On Day 8, the patients will start maintenance treatment of 300 mg BID for the duration of the treatment period.
  Arms: AZD3241, 300 mg
Drug: AZD3241 600 mg BID — The following dose escalation schedule will be used for 600 mg BID: 100 mg BID from Day 1 through Day 7 and 300 mg BID from Day 8 through Day 14. On Day 15, the patients will start maintenance treatment of 600 mg BID for the duration of the treatment period.
  Arms: AZD3241, 600 mg
Drug: Placebo — Placebo to AZD3241 BID
  Arms: Placebo

SUMMARY:
This is a study where AZD3241 or placebo is given to patients with Parkinson's disease in a blinded and randomized assignment. The main objective is to see if safety and tolerability of the drug is acceptable.

DETAILED DESCRIPTION:
A Phase IIa, 12 Week, Multicentre, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group Study to Assess the Safety and Tolerability of Oral AZD3241 in Patients with Parkinson's Disease

ELIGIBILITY:
Inclusion Criteria:

* Each patient must be able and willing to provide signed and dated informed consent prior to the study.
* Female and male patients aged 30 to 80 years at the day of enrollment (Visit 1).
* Patients must meet the criteria for "Diagnosis of idiopathic Parkinson's disease" according to the UKPDS Brain Bank criteria (Hughes et al 1992).
* Have a modified Hoehn and Yahr stage 1-2.5.
* Having no treatment for Parkinson's disease and have no need to add anti-Parkinson's disease treatment during the 14 weeks of study OR are on stable anti-Parkinson's disease medication.

Exclusion Criteria:

* Diagnosis is unclear or a suspicion of other Parkinsonian syndromes exists, such as secondary Parkinsonism (caused by drugs, toxins, infectious agents, vascular disease, trauma, brain neoplasm), Parkinson-plus syndromes or heredodegenerative diseases.
* Have undergone surgery for the treatment of Parkinson's disease (eg, pallidotomy, deep brain stimulation, fetal tissue transplantation) or have undergone any other brain surgery at any time, even for non-Parkinson's disease conditions.
* Presence of dyskinesias, motor fluctuations, swallowing difficulties or loss of postural reflexes, defined as scoring 2 or more on item 30 of the UPDRS.
* Current/history of psychiatric diagnosis of acute psychotic disorder or other primary psychiatric diagnoses, i.e. bipolar disorder or MDD, or other psychiatric, neurological or behavioral disorders/symptoms that may interfere with conduct of study.
* Current significant major or unstable respiratory disease, heart disease, cerebrovascular disease, hematological disease, hepatic disease, renal disease, gastrointestinal (GI) disease, or other major disease as judged by the investigator.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2012-10; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Change from baseline in vital signs. | Screening (baseline), randomization, after 2, 4, 8 and 12 weeks of treatment and 2 weeks after termination of treatment (week 14)
  Vital signs: systolic and diastolic blood pressure and pulse including orthostatic challenge will be assessed. Change from baseline at each visit will be calculated as the visit value minus the baseline value for each vital sign: Blood Pressure, pulse rate (supine and standing), weight and oral temperature.
Change from baseline in Physical Exam results. | Baseline and 2 weeks after termination of treatment (week 14)
  Assessment of general appearance, skin, head and neck, lymph nodes, thyroid, abdomen, cardiovascular, respiratory, and neurological systems, including full palpation of thyroid gland.
Change from baseline in Suicidality as assessed by the Columbia-Suicide Severity Rating Scale (CSSRS). | screening (baseline), randomization, after 2, 4, 8 and 12 weeks of treatment and 2 weeks after termination of treatment (week 14)
  Suicidality as assessed by the Columbia-Suicide Severity Rating Scale (CSSRS) The CSSRS assesses the suicidal behavior and suicidal ideation in patients. Occurrence of suicidal behavior is defined as having answered "yes" to a least 1 of the 4 suicidal behavior sub categories (actual attempt, interrupted attempt, aborted attempt, and preparatory acts or behavior) at any post randomization evaluation. Occurrence of suicidal ideation after randomization is defined as having answered "yes" to at least one of the suicidal ideation sub-categories (wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods [not plan] without intent to act, active suicidal ideation with some intent to act [without specific plan], and active suicidal ideation with specific plan and intent) at any post randomization evaluation.
Adverse events (AEs) including frequency and severity. | Screening, randomization, week 1, 2, 4, 8, 12, 14
Change from baseline in laboratory safety assessments. | Screening (baseline), randomization, after 2, 4, 8 and 12 weeks of treatment and 2 weeks after termination of treatment (week 14)
  Change from baseline at each visit will be calculated as the visit value minus the baseline value for each continuous clinical chemistry, hematology and urinalysis measurements.
  Abnormal or out-of-range values will be flagged.
Change from baseline in 12-lead ECG. | Screening (baseline), randomization, after 2, 4, 8 and 12 weeks of treatment and 2 weeks after termination of treatment (week 14)
  Change from baseline at each visit will be calculated as the visit value minus the baseline value for each ECG parameter: heart rate, QRS duration, PR interval, RR interval, QT and calculated QTcF interval. Abnormal or out-of-range values will be flagged.

SECONDARY OUTCOMES:
Pharmacokinetics (PK) of AZD3241 in the terms of Cmax, Cmin, and AUC0-t. | Randomization and after week 1, 2, 4, 8, and 12 weeks of treatment
  Blood samples (5 mL) for determination of AZD3241 concentration in plasma will be collected in accordance with the information in the Study Plan. PK analysis will be based on the PK analysis set. Plasma concentrations of AZD3241 will be determined and PK analyzed by a population PK model.
  PK analysis will be based on the PK analysis set and will include determination of observed Cmax, Cmin, and AUC0-t. Plasma drug concentrations of AZD3241 will be determined and PK analyzed by a population PK model. If the quality of the data does not allow a population PK analysis, plasma concentrations from all patients will be analyzed graphically and by descriptive statistics, as appropriate.
Pharmacodynamic effect of AZD3241 in the terms of Myeloperoxidase (MPO) activity in plasma. | Screening (baseline), randomization, after, 4, 8 and 12 weeks of treatment and 2 weeks after termination of treatment (week 14)

CONTACTS AND LOCATIONS:
Overall Officials: Joel Posener, MSD, Study Director — AZ Neuro
Locations (13):
- United States (13):
  - Research Site, Birmingham, Alabama
  - Research Site, Long Beach, California
  - Research Site, New Haven, Connecticut
  - Research Site, Atlantis, Florida
  - Research Site, Boca Raton, Florida
  - Research Site, Orlando, Florida
  - Research Site, Sunrise, Florida
  - Research Site, Tampa, Florida
  - Research Site, Kansas City, Kansas
  - Research Site, Bingham Farms, Michigan
  - Research Site, Omaha, Nebraska
  - Research Site, Lawrenceville, New Jersey
  - Research Site, Marlton, New Jersey